CLINICAL TRIAL: NCT06813404
Title: Building Strength for Menopause
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfunded
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB# 24-12-12
Record Dates: First submitted 2025-01-27; First posted 2025-02-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Strength Training Effects; Menopausal Women; Cognitive Function
Keywords: menopausal women, strength training, cognitive function
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Feasibility pilot study of heavy resistance training for middle-aged, menopausal women.
Who Masked: Outcomes Assessor
Masking Description: Data analysis will be blinded such that the analyst does not know which group each result is associated with. Efforts will be made to have final testing blinded, however if resources are limited, final testing will be done by exercise intervention leads.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First wave of participants (n=30) (Experimental): This arm is the first round of the exercise intervention, conducted with half (n=30) the anticipated number of participants.
  Interventions: Behavioral: Heavy resistance training; Behavioral: Yoga
- Second wave of participants (n=30) (Experimental): This arm is the second round of participants (n=30) who will receive the same intervention as the first wave.
  Interventions: Behavioral: Heavy resistance training; Behavioral: Yoga

INTERVENTIONS:
Behavioral: Heavy resistance training — The heavy resistance training intervention will consist of twice weekly exercise sessions of 60 minutes each.
Behavioral: Yoga — Twice weekly yoga sessions of 60 minutes each

SUMMARY:
A pilot study investigating whether heavy resistance training is enjoyable, acceptable, and feasible for middle-aged women undergoing the menopausal transition. Additional outcomes to be assessed include changes to strength and muscle composition as well as changes to cognitive function and self-reported measures of fatigue, cognition, self-efficacy, and mood.

ELIGIBILITY:
Inclusion Criteria:

* 40-60 years of age at study enrollment
* Currently experiencing symptoms related to menopause
* Low physical activity levels at study enrollment (not meeting CDC guidelines of 150 minutes moderate/75 minutes vigorous activity per week)
* No regular (>1x per week) participation in heavy resistance training or yoga exercise within the past 6 months
* Physician's consent to participate in strength testing and the exercise program (if deemed necessary)
* Ambulatory
* Absence of health conditions that may be exacerbated by exercise
* Good or corrected vision and hearing
* Intention to remain in the Boston area for the duration of the study
* Willingness to complete study assessments
* Ability to read, write and understand English
* Not currently enrolled in another PA study

Exclusion Criteria:

* Under 40 or over 60 years
* Pregnant or planning to become pregnant
* Moderate to high physical activity levels at enrollment (meeting CDC guidelines)
* Currently participating regularly (>1x per week) in a heavy resistance training or yoga program
* Non-consent of physician (if deemed necessary)
* Non-ambulatory (e.g. use of walkers, wheelchairs)
* Presence of health conditions that may be exacerbated by exercise (arthritis, musculoskeletal disorders, etc.)
* Problems with vision or hearing
* Intent to move or take an extended (>2 weeks) vacation during the testing time points (baseline, 4 months)
* Unwilling to complete study assessments
* Currently enrolled in another PA study

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility (adherence) | From enrollment to the end of the exercise intervention at 16 weeks
  Adherence to the study intervention will be evaluated at the end of each arm, based on recorded attendance. It will be recounted as a percentage.
Feasibility (retention) | From enrollment to the end of the exercise intervention at 16 weeks
  Retention of participants in each group will be evaluated at the end of each arm, based on recorded attendance. It will be recounted as a percentage.
Acceptability | From enrollment to the end of the exercise intervention at 16 weeks
  Participant enjoyment will be evaluated at the end of each arm, based on self-reported enjoyment after each session, and a final survey for participant feedback on the intervention. Enjoyment will be rated on a Likert scale.

SECONDARY OUTCOMES:
Muscular strength | From baseline testing to the end of the exercise intervention at 16 weeks
  Assessed through 1-repetition maximum testing of two compound lifts: barbell box squat and barbell bench press. Tests will be conducted at baseline and at the end of the intervention for both exercise groups.
Cognitive function (executive function) | From baseline testing to the end of the exercise intervention at 16 weeks
  The Digit Symbol Substitution test will be used to assess components of executive function such as processing speed, working memory, visuospatial processing, and attention. This is recorded as total number of trials and total number of correct trials in 90 seconds.
Cognitive function (working memory) | From baseline testing to the end of the exercise intervention at 16 weeks
  The Backward Digit Span test will be used to assess working memory and attention. This test is scored as the longest sequenced reached and passed and the total number of attempts.
Cognitive function (memory recall) | From baseline testing to the end of the exercise intervention at 16 weeks
  The East Boston Memory Test will be used to assess immediate and delayed recall. The test is scored as the correct number of components recalled from a three-sentence story.

OTHER OUTCOMES:
Body composition | From baseline testing to the end of the exercise intervention at 16 weeks
  As an option, participants may complete a DEXA scan to assess body composition. This will be used to assess changes to lean body mass.

CONTACTS AND LOCATIONS:
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data will be de-identified